CLINICAL TRIAL: NCT04598828
Title: Using Time Varying Non-Invasive Neuromodulation to Improve Neurovascular Status in Parkinson's Disease
Brief Title: Use of a Non-Invasive Brainstem Neuromodulation Device to Improve Neurovascular Status in Parkinson's Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of activity and not meeting recruitment goals within expected timeframe
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00067408
Record Dates: First submitted 2020-10-16; First posted 2020-10-22 (Actual); Results first posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-06

CONDITIONS: Parkinson Disease
Keywords: balance disorders; motor functions
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Treatment 1 (Experimental): Participants will receive Experimental treatment 1 stimulation for a duration of 12 weeks, twice daily for 19 minutes
  Interventions: Device: Non-invasive brainstem stimulation
- Treatment 2 (Experimental): Participants will receive Experimental treatment 2 stimulation for a duration of 12 weeks, twice daily for 19 minutes
  Interventions: Device: Non-invasive brainstem stimulation

INTERVENTIONS:
Device: Non-invasive brainstem stimulation — Study participants will self-administer ~19-minute treatments twice daily in the home setting using a non-invasive brainstem modulation device. The device has been deemed as a nonsignificant risk for studies in Parkinson's disease by the United States Food and Drug Administration.

SUMMARY:
This study is a single-site, double-blinded, randomized clinical trial designed to elucidate mechanism(s) of action for symptomatic benefits observed in Parkinson's disease (PD)

DETAILED DESCRIPTION:
Patients treating twice daily using a non-invasive brainstem modulation device. Study participants will self-administer treatments in the home setting over a period of 12 weeks. Changes in cerebral blood flow perfusion, cerebrovascular reactivity and functional connectivity between the pre-treatment baseline and the end of the treatment period will be monitored and compared to changes in validated standardized clinical measures of motor and non-motor symptoms in PD.

ELIGIBILITY:
Inclusion Criteria:

* Must be 21-85 years old
* Diagnosed with Parkinson's Disease
* Within driving distance of Atrium Health Wake Forest Baptist (Winston-Salem, NC)
* Responsive to Parkinson's medication for a minimum of 3 years
* Have ability to reliably use the investigational device
* Understand and complete all assessments (provided in English only)
* Be able to have 3 separate MRI scans (1.5 hours per MRI)
* Have a study partner/regular caregiver that is willing to participate in the trial
* Demonstrate moderate burden of motor symptoms and non-motor symptoms
* Consent to being videotaped during motor examination visit
* Willing to answer questions related to sexual interest, arousal and performance in an interview with study staff

Exclusion Criteria:

* Cannot attend all study visits (4 on-site visits) or complete all study activities
* Heart attack, angina, or stroke within the past year
* Use medications that regulate heart rate
* Have a history or prior diagnosis of dementia
* Receiving deep brain stimulation therapy
* Treated with a pump for continuous delivery of dopamine replacement therapy
* Use of Apomorphine rescue
* Works night shifts
* Have any significant co-morbidity such as stroke, brain tumor, epilepsy, Alzheimer's disease, multiple sclerosis, ALS, atypical Parkinsonism, or aneurysm
* History or evidence of unstable mood disorder or demonstrates evidence of suicidality
* Hearing aids that are implanted or cannot be easily removed and replaced, such as cochlear implants
* Chronic ringing in the ears for more than 3 months
* Diagnosed with traumatic brain injury with ongoing symptoms
* Recent history of substance abuse and/or dependence (alcohol or other drugs)
* Diagnosed balance dysfunction
* Eye surgery within the previous 3 months
* Ear surgery within the previous 6 months
* Active ear infection, perforated tympanic membrane, or inner ear inflammation
* Recent history of frequent ear infections (≥ 1 per year over the past two years)
* Contraindications for MRI scans, such as metal implants or a pacemaker
* Currently enrolled or have participated in another interventional clinical trial within the last 30 days
* Taking medication for vomiting or nausea more than 2 times per week, consistently
* Ongoing symptoms from a COVID-19 infection that includes one or more of the exclusion criteria listed above
* Planned surgery scheduled to occur during the clinical trial that requires sedation and/or would typically be followed with a prescription for pain management
* Women who are pregnant or plan to become pregnant during the the study

Women of child-bearing potential (i.e., are not yet 3 years removed from their first menopausal symptom), who are not abstinent or exclusively in same sex relationships must:

Test negative for pregnancy as indicated by a negative urine pregnancy test

Agree to use an approved contraception method

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-07-06 (Actual); Primary Completion 2023-10-02 (Actual); Study Completion 2024-10-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher T Whitlow, MD, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be available to other researchers.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment 1 | Treatment 2
Started | 6 | 6
Completed | 5 | 4
Not Completed | 1 | 2
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment 1 | Treatment 2 | Total
Number analyzed (Participants) | 5 | 4 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 3 | 3 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.2 (9.20) | 68.5 (2.52) | 70.6 (6.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 4 | 9
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 4 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Cerebral Blood Flow (CBF) Perfusion
Description: Cerebral blood flow (CBF) measured using pseudo Continuous Arterial Spin Labeling (pCASL) magnetic resonance imaging (MRI) will be used to monitor changes in global perfusion
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: ml/100g/min
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 5 | 4
ml/100g/min | 35.5 (4.76) | 35.2 (5.94)

2. Primary Outcome: Cerebral Blood Flow (CBF) Perfusion
Description: as for outcome 1
Time Frame: end of treatment (week 12)
Measure: Mean (Standard Deviation); unit: ml/100g/min
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 5 | 4
ml/100g/min | 33.6 (3.77) | 33.3 (10.38)

3. Primary Outcome: Cerebrovascular Reactivity
Description: Cerebral blood flow is measured with pCASL MRI at baseline and during hypercapnic challenge. The percent change in CBF is divided by the increase in end-tidal CO2 measured in mmHg, measured with RespirACT system
Time Frame: baseline
Population: Only 3 total participants had usable data
Measure: Mean (Standard Deviation); unit: % change CBF/change in CO2 (mmHg)
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 1 | 2
% change CBF/change in CO2 (mmHg) | 1.01 (NA) — For N=1, there is no SD value. | -1.39 (1.57)

4. Primary Outcome: Cerebrovascular Reactivity
Description: as for outcome 3
Time Frame: end of treatment (week 12)
Population: Only 3 total participants had usable data
Measure: Mean (Standard Deviation); unit: % change CBF/change in CO2 (mmHg)
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 1 | 2
% change CBF/change in CO2 (mmHg) | -1.94 (NA) — For N=1, there is no SD value. | -0.7 (0.96)

5. Secondary Outcome: Percent Change in Functional Connectivity
Description: Changes to the within-network connectivity of the DMN (Default Mode Network)
Time Frame: baseline and end of treatment (week 12)
Measure: Mean (Standard Deviation); unit: Percent Change in Default Mode Network
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 5 | 4
Percent Change in Default Mode Network | 1.1 (21.8) | 7.5 (19.2)

6. Other Pre Specified Outcome: Change in Cerebral Haemodynamics
Description: Transcranial Doppler sonography (TCD), a non-invasive ultrasound, will be used to monitor changes in cerebral blood flow velocity (cm/s) in response to a hypercapnic challenge.
Time Frame: baseline and end of treatment (week 12)
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Durability of Change of Cerebral Blood Flow (CBF) Perfusion
Description: Arterial arrival time (AAT) measured using pseudo Continuous Arterial Spin Labeling (pCASL) magnetic resonance imaging (MRI) will be used to monitor changes in global perfusion.
Time Frame: baseline and the post-treatment follow-up (week 17)
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Durability of Change of Cerebrovascular Reactivity
Description: AAT measured using pCASL MRI after a hypercapnic challenge will be used to monitor changes in cerebrovascular reactivity
Time Frame: baseline and the post-treatment follow-up (week 17)
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Durability of Change of Functional Connectivity
Description: Resting-state magnetic resonance imaging (rs-MRI) will be used to monitor changes in functional connectivity
Time Frame: baseline and the post-treatment follow-up (week 17)
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Change in the Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS)
Description: Used to follow the longitudinal course of symptoms of Parkinson's disease - Each parkinsonian sign or symptom is rated on a 5-point Likert-type scale (ranging from 0 to 4), with higher scores indicating more severe impairment. The maximum total UPDRS score is 199, indicating the worst possible disability from PD
Time Frame: baseline, end of treatment (week 12), and the post-treatment follow-up (week 17)
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Change in the Timed Up and Go Test
Description: To determine fall risk and measure the progress of balance, sit to stand and walking (ranging from ≤10 seconds as normal to 30 seconds as high fall risk).
Time Frame: baseline, end of treatment (week 12) and the post-treatment follow-up (week 17)
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Change in the Montreal Cognitive Assessment
Description: Cognitive screening test - range from zero to 30, with a score of 26 and higher generally considered normal.
Time Frame: baseline, end of treatment (week 12) and the post-treatment follow-up (week 17)
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Change in the Non-Motor Symptom Scale
Description: Scale to assess a wide range of non-motor symptoms in patients with Parkinson's disease - 30-item rater-based scale to assess a wide range of non-motor symptoms in patients with Parkinson's disease (PD). The Non-Motor Symptom Scale measures the severity and frequency of non-motor symptoms across nine dimensions - the total score significantly increased with disease severity and duration meaning that the number of individual non-motor symptoms reported by our patients increases as the disease progresses. Score range 0 - 360.
Time Frame: Change between the baseline and end of treatment (week 12) measure.
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Change in the Non-Motor Symptom Scale
Description: as for outcome 13
Time Frame: Change between the baseline and the post-treatment follow-up (week 17) measure.
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Change in the Geriatric Depression Scale
Description: A self-report measure of depression in older adults - Scores of 0-4 are considered normal, depending on age, education, and complaints; 5-8 indicate mild depression; 9-11 indicate moderate depression; and 12-15 indicate severe depression.
Time Frame: baseline, end of treatment (week 12) and the post-treatment follow-up (week 17)
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Change in the Parkinson's Anxiety Scale
Description: Anxiety assessment - The PAS is a 12-item observer or patient-rated scale with three subscales, for persistent, episodic anxiety and avoidance behavior - There is a maximum total score of 48. Higher scores indicate great experiences of anxiety.
Time Frame: baseline, end of treatment (week 12) and the post-treatment follow-up (week 17)
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Change in the Epworth Sleepiness Scale
Description: A self-administered questionnaire to assess the daytime sleepiness - The ESS score (the sum of 8 item scores, 0-3) can range from 0 to 24. The higher the ESS score, the higher that person's average sleep propensity in daily life (ASP), or their 'daytime sleepiness'.
Time Frame: baseline, end of treatment (week 12) and the post-treatment follow-up (week 17)
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Change in the Functional Assessment of Chronic Illness Therapy - Fatigue
Description: A tool to help manage chronic illness - The responses to the 13 items on the FACIT fatigue questionnaire are each measured on a 4-point Likert scale. Thus, the total score ranges from 0 to 52. High scores represent less fatigue
Time Frame: baseline, end of treatment (week 12) and the post-treatment follow-up (week 17)
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Change in Arterial Stiffness
Description: Arterial stiffness will be assessed as carotid-femoral pulse wave velocity (PWV). PWV is calculated by dividing the distance between the carotid and femoral arteries by the pulse transit time.
Time Frame: baseline and end of treatment (week 12)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 17 weeks
Description: Treatment site discomfort, Headache, Ear pain, Tinnitus
Arm/Group | Treatment 1 | Treatment 2
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4
Other Adverse Events (participants affected / at risk) | 5/5 | 2/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment 1 (N=5) | Treatment 2 (N=4)
Treatment site discomfort (General disorders) | 4 (4) | 0 (0)
Tinnitus (General disorders) | 1 (1) | 0 (0)
Headache (General disorders) | 0 (0) | 1 (1)
Ear pain (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-07-24): https://cdn.clinicaltrials.gov/large-docs/28/NCT04598828/Prot_SAP_000.pdf
  • Informed Consent Form (2024-06-27): https://cdn.clinicaltrials.gov/large-docs/28/NCT04598828/ICF_001.pdf